CLINICAL TRIAL: NCT02817711
Title: Lyon BJI Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0388
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Bone and Joint Infection
Keywords: infection; bone and joint infection; relapse; adverse event
MeSH Terms: conditions — Infections; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prospective Cohort includes all patients with bone or joint infection (BJI), with or without implant. The aim of this Cohort is to improve the knowledges about the treatment failure and the occurrence of serious adverse events. Various data of patients included are collected and will be analysed.

Patients with a bone or joint infection are treated at the department of infectious diseases, at Infectious disease department of Hospices Civils de Lyon. They have regularly a consultation with a physician: 2-3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery and 24 months after surgery. It allows to the physician to follow the evolution of the patient under treatment and after discontinuation of the treatment.

Several data are collected during the follow-up concerning: demographics data, treatment including the use of off-label antibiotics for the treatment of BJI, adverse events, microbiology, surgeries, healing or relapse, date of symptoms, ASA score, implant or not. If there is an implant, the date of implantation and the number of the prosthesis infected are collected.

This cohort allows to improve knowledge concerning the treatment failure and the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients with bone or joint infection, with or without implant

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes all patients who have a bone and joint infection, with or without implant, and treated in the department of infectious disease at the HCL.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2002-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Treatment Failure in patients with bone or joint infection | 2 years
  Up to 30% of patients experience a relapse, even when the treatment is considered as optimal. This Cohort will improve knowledges about the mechanisms of treatment failure by collecting data concerning infectious disease, surgery and microbiology and by analysing the cases where treatment failed. Treatment failure is defined by local clinical and/or microbiological relapse, under treatment or after treatment discontinuation.

SECONDARY OUTCOMES:
Occurrence of serious adverse events in patients with bone or joint infection | 6 months
  The duration of the antibiotic treatment is long : several weeks, several months or even several years in some cases. Patients are then exposed to adverse events. The data concerning theses adverse events are collected in this Cohort : molecule, dosage, description of the adverse event, a change in treatment. A severity grade is allocated to every adverse event, based on the " Common Terminology Criteria for Adverse Events ". This is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term (from 1 to 5). Severe adverse events have a grade >=3.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, MD, PhD, Principal Investigator — Centre de reference des infections ostéo-articulaires
Locations (1):
- Centre de reference des infections ostéo-articulaires, Hôpital de la Croix-Rousse, 103 Grande Rue de la Croix-Rousse, Lyon, France

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr/